CLINICAL TRIAL: NCT05568472
Title: A Randomized Phase III Trial Comparing Active Symptom Monitoring Plus Patient Education Versus Patient Education Alone to Improve Persistence With Endocrine Therapy in Young Women With Stage I-III Breast Cancer (ASPEN)
Brief Title: Monitoring Symptoms to Help Young Women Take Hormone Therapy for Stage I-III Breast Cancer, ASPEN Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: S2010; NCI-2022-06902 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2010 (Other: SWOG); SWOG-S2010 (Other: DCP); S2010 (Other: CTEP); R01CA266012 (NIH); UG1CA189974 (NIH)
Record Dates: First submitted 2022-09-23; First posted 2022-10-05 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Hormone Receptor-Positive Breast Carcinoma
MeSH Terms: interventions — Practice Guidelines as Topic; Standard of Care; Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM I (ET, health education, symptom assessment) (Experimental): Patients receive ET and standard of care clinic visits with a cancer provider at 12, 24, 36, 48, 60, and 72 weeks, and phone visit at 80 weeks to access ongoing use ET medication. Patients are asked 6 brief questions about symptoms weekly by email, text, or phone call for the first 6 months, then every 4 weeks for 12 months. Patients also receive a list of websites with information about breast cancer, side effects of breast cancer medicines, and ways to help with heart health. Patients have the option to submit blood specimen collection at baseline, 3, 12, and 18 months.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Procedure: Endocrine Drug Therapy; Behavioral: Health Education; Other: Questionnaire Administration; Other: Symptom Specific Assessment Tool
- ARM II (ET, health education) (Active Comparator): Patients receive ET and standard of care clinic visits with a cancer provider at 12, 24, 36, 48, 60, and 72 weeks, and phone visit at 80 weeks to access ongoing use ET medication. Patients also receive a list of websites with information about breast cancer, side effects of breast cancer medicines, and ways to help with heart health. Patients have the option to submit blood specimen collection at 3, 12, and 18 months.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Procedure: Endocrine Drug Therapy; Behavioral: Health Education; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Standard of care hormone therapy and standard visit with clinician
  Other Names: standard of care; standard therapy
Procedure: Biospecimen Collection — Undergo correlative studies
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Endocrine Drug Therapy — Undergo endocrine therapy
Behavioral: Health Education — Receive list of websites
Other: Questionnaire Administration — Ancillary studies
Other: Symptom Specific Assessment Tool — Receive a weblink via email or text message and asked 6 brief questions about symptoms
  Other Names: Symptom Assessment Tool; Symptom-Specific Assessment Tool
  Arms: ARM I (ET, health education, symptom assessment)

SUMMARY:
This phase III trial compares the effect of active symptom monitoring and patient education to patient education alone in helping young women with stage I-III breast cancer stay on their hormone therapy medicines. The patient education tool contains interactive weblinks which provide patients with education material about breast cancer and side effects of therapy. Symptom monitoring is a weblink via email or text message with questions asking about symptoms. Hormone therapy for breast cancer can cause side effects, and may cause some women to stop treatment early. Asking about symptoms more often may help women keep taking hormone therapy medicines.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare persistence with the initially prescribed oral endocrine therapy (ET) through 72 weeks for young women being treated for hormone-receptor positive stage I-III breast cancer randomized to Active Symptom Monitoring (ASM) + patient education or patient education alone.

SECONDARY OBJECTIVES:

I. To compare patient-reported adherence with the initially prescribed oral ET over time as assessed with the Voils measure between the two arms.

II. To compare worst pain as assessed with the Brief Pain Inventory, in aromatase inhibitors-treated (AI-treated) participants over time between the two arms.

III. To compare hot flashes as assessed with the Functional Assessment of Cancer Therapy-Endocrine Symptoms (FACT-ES) Endocrine Symptoms Scale in tamoxifen-treated participants over time between the two arms.

EXPLORATORY OBJECTIVES:

I. To describe key treatment-emergent symptoms as assessed with the Brief Pain Inventory, the Patient-Reported Outcomes Measurement Information System (PROMIS-29) Profile, the PROMIS Cognitive Function, and the FACT-ES Endocrine Symptoms Scale over time between the two arms.

II. To develop a composite risk prediction model (including demographics, socioeconomic variables, and clinical variables) to identify participants who are most likely to benefit from ASM.

III. To examine associations between baseline symptom bother as assessed with the GP5 item from the FACT-ES and persistence with oral ET.

IV. To examine the pattern by arm of treatment toxicity from the oral ET agents that are prescribed in this study over time during the first 24 weeks.

V. To compare biochemically determined adherence with the initially prescribed oral ET as assessed with centrally evaluated drug concentrations and metabolites between ASM + patient education and patient education alone over time.

VI. To examine associations overall and by arm between baseline estradiol concentrations evaluated centrally and development of treatment-emergent symptoms as assessed with the Brief Pain Inventory, the PROMIS-29 Profile, the PROMIS Cognitive Function, and the FACT-ES endocrine symptoms scale.

VII. To determine patterns of change overall and by arm in centrally evaluated estradiol concentrations during study participation in participants with chemotherapy-induced ovarian failure, those receiving gonadotrophin releasing hormone (GnRH) agonist therapy, and those who had undergone bilateral salpingo-oophorectomy.

VIII: To identify inherited genetic variants using genome-wide genotyping that contribute to development of endocrine therapy-emergent toxicity.

BANKING OBJECTIVE:

I. To bank specimens for future correlative studies.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive ET and standard of care clinic visits with a cancer provider at 12, 24, 36, 48, 60, and 72 weeks, and phone visit at 80 weeks to access ongoing use ET medication. Patients are asked 6 brief questions about symptoms weekly by email, text, or phone call for the first 6 months, then every 4 weeks for 12 months. Patients also receive a list of websites with information about breast cancer, side effects of breast cancer medicines, and ways to help with heart health. Patients have the option to submit blood specimen collection at baseline, 3, 12, and 18 months.

ARM II: Patients receive ET and standard of care clinic visits with a cancer provider at 12, 24, 36, 48, 60, and 72 weeks, and phone visit at 80 weeks to access ongoing use ET medication. Patients also receive a list of websites with information about breast cancer, side effects of breast cancer medicines, and ways to help with heart health. Patients have the option to submit blood specimen collection at 3, 12, and 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be female and have Stage I, II, or III hormone receptor positive breast cancer based on clinical or pathologic evaluation
* Participants must have been pre- or peri-menopausal at the time of breast cancer diagnosis by satisfying one of the following:

  * had a menstrual period (by self-report) within the 12 months before breast cancer diagnosis, or
  * had a serum or plasma estradiol and/or follicle stimulating hormone (FSH) concentration consistent with premenopausal status (based on institutional standards) within the 12 months before breast cancer diagnosis or when checked after breast cancer diagnosis
* Participants must have started initial treatment with standard of care oral endocrine therapy (ET) (i.e., tamoxifen, anastrozole, exemestane, or letrozole; within 14 days prior to randomization or be planning to start initial treatment with standard of care oral ET within 14 days after randomization
* Participants who currently have ovarian function (estradiol above the postmenopausal range) must be planning to undergo ovarian suppression or ablation concomitantly with oral ET medication, starting before or at the same time as oral ET initiation. Participants with chemotherapy-induced amenorrhea or ovarian failure at time of registration must be planning to start ovarian suppression or ablation if they have recurrence of ovarian function during study participation (circulating estradiol concentration in the premenopausal range or recurrence of menses)
* Participants must have completed surgery for treatment of breast cancer at least 14 days prior to randomization NOTE: Concomitant radiotherapy at the time of randomization and/or during study participation is allowed
* Participants who received chemotherapy must have finished it at least 14 days prior to randomization NOTE: Concomitant maintenance targeted or biologic therapy (e.g., human epidermal growth factor receptor 2 [anti-HER2] therapy, poly-ADP ribose polymerase [PARP] inhibitor therapy, CDK4/6 inhibitor therapy, osteoclast inhibitor therapy) at the time of randomization and/or during study participation is allowed
* Participants must be >= 18 years of age
* Participants must have a complete medical history within 60 days prior to randomization
* Participants must be able to complete Patient-Reported Outcome (PRO) instruments in English or Spanish

Participants must:

* agree to complete PROs at all scheduled assessments and
* complete the pre-registration (baseline) PRO forms within 14 days prior to randomization

  * Participants must be able to complete symptom questions on a web browser (on a smartphone, tablet, or computer) or respond via voice on a telephone in English or Spanish. Participants must agree to complete symptom questions at all scheduled assessments NOTE: Participants who do not have access to the internet and who cannot receive telephone calls for interactive voice response system (IVRS) assessments are not eligible
  * Participants must be offered the opportunity to participate in specimen banking for translational medicine. With participant consent, specimens must be collected and submitted via the Southwest Oncology Group (SWOG) specimen tracking system
  * Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines

Exclusion Criteria:

* Participants must not have distant metastatic breast cancer
* Participants who have started or plan to start treatment with tamoxifen during study participation must not have received prior tamoxifen for treatment or prevention of breast cancer
* Participants who have started or plan to start treatment with an aromatase inhibitor during study participation must not have received prior aromatase inhibitor therapy for treatment or prevention of breast cancer
* Participants must not be taking or planning to take oral estrogen-or progesterone-containing treatments during study participation

NOTES:

* Participants who start or plan to start treatment with an aromatase inhibitor may have previously received tamoxifen for prevention of breast cancer or treatment of a prior cancer
* Participants may have received prior treatment with an aromatase inhibitor for infertility treatment
* Participants must not be planning to become pregnant during the 80 weeks of study participation

  * Participants must not receive additional anti-cancer treatments (i.e., experimental therapy, immunotherapy, biologics, etc.) as part of another clinical trial
  * Participants must not have a non-breast malignancy for which they are currently receiving treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 565 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Persistence with initially prescribed oral estrogen (ET) medication | From randomization to discontinuation of the initially prescribed ET for more than 60 days or switching to a new oral ET medication, assessed up to 72 weeks
  Will be assessed by the treating provider at each study visit every 12 weeks and prospectively documented on the S2010 treatment log, including any switch from the initially prescribed oral ET. Persistence with initially prescribed oral ET by intervention arm out to 72 weeks will be described using Kaplan-Meier plots. Potential differences by arm will be tested using multivariable Cox regression. Persistence with any oral ET (aromatase inhibitor [AI] and/or tamoxifen) at 72 weeks by arm will be examined in a consistent manner. The study stratification variables (age [< 45 vs >= 45], chemotherapy [yes/no], and ET [AI vs tamoxifen]), as well as race, ethnicity, and disease stage, will be included as covariates in the regression models. In the timeframe of evaluation, censored events (newly diagnosed cancer, cancer recurrence, or death) are anticipated to be low.

SECONDARY OUTCOMES:
Occurrence of any non-adherence | Up to 18 months
  Will be assessed using the Voils validated adherence tool that both determines the extent of nonadherence as well as reasons for non-adherence. Kaplan Meier plots will be used to describe patterns of non-adherence between arms. Multivariable Cox regression will be used to assess this secondary endpoint.
Worst pain | Up to 12 weeks
  Will be measured using the Brief Pain Inventory - Short Form (BPI-SF) "worst pain" question ("Please rate your pain by circling the one number that best describes your pain at its worst in the last 24 hours") in the subset of patients planning to receive AI treatment. Worst pain is measured on an 11-point scale of 0 ("no pain") to 10 ("pain as bad as you can imagine"). Linear regression will be used, adjusting for the stratification factors and the baseline score.
Incidence of hot flashes | Up to 12 weeks
  Will be assessed using the Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES) "I have hot flashes/hot flushes" (ES1) question in the subset of patients planning to receive tamoxifen therapy. Hot flashes/hot flushes are measured on a scale of 0 ("not at all") to 4 ("very much"), with higher values indicating increased concern over the past 7 days. Linear regression will be used to compare scores between arms, adjusting for the stratification factors and the baseline score.

OTHER OUTCOMES:
Symptom bother | Up to 18 months
  Assessed using the Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES) "I am bothered by side effects of treatment" (GP5) question. This is rated on a scale of 0 ("not at all") to 4 ("very much") with higher values indicating worse physical well-being over the past 7 days.
Symptom burden: average pain | Up to 18 months
  Will be measured using the Brief Pain Inventory - Short Form (BPI-SF) average pain question "Please rate your pain by marking the box beside the number that best describes your pain on the average", range 0 to 10, with 0 representing "no pain" and 10 representing "pain as bad as you can imagine."
Symptom burden: pain interference | Up to 18 months
  Will be measured using the Brief Pain Inventory - Short Form (BPI-SF) pain interference scale, range 0 to 10, with lower values representing "no interference" and 10 signifying "complete interference."
Symptom burden: overall health profile | Up to 18 months
  Will be measured using the Patient-Reported Outcomes Measurement Information System 29 (PROMIS-29) profile subscales: fatigue (33-76), sleep disturbance (32-74), physical function (22-57), depression (41-80), anxiety (40-82), and ability to participate in social roles and activities (27-65). Raw scores (range 4-20 for all subscales) are converted to T scores (approximate ranges shown next to subscale), with mean 50 and standard deviation 10. The T score conversion is handled programmatically by Health Measures and depends upon the number of questions answered, minimums and maximums may differ from those shown here. Higher T scores represent more of the characteristic being measured (e.g., higher T score on fatigue score represents more fatigue, but higher T score on physical function represents better physical function).
Symptom burden: cognitive function | Up to 18 months
  Will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Cognitive Function 4a. Raw scores (range 4 to 20) are converted to a T score with mean 50, and standard deviation 10. The approximate minimum and maximum T scores for this scale are 24 and 62 respectively, with higher T scores representing better cognitive function. T score conversion is handled programmatically by Health Measures and depends upon the number of questions answered; actual minimums and maximums may differ depending upon the number of questions answered.
Symptom burden: endocrine symptoms | Up to 18 months
  Will be measured using the Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES) Endocrine Symptoms Scale. This is a 19-item subscale with range 0 to 76, with higher values representing better quality of life.
Estradiol concentration | Up to 18 months
  Plasma concentrations of estradiol will be quantitated centrally using a tandem mass spectroscopy-based ultrasensitive estradiol assay
Adherence to medications based on plasma concentrations | Up to 18 months
  Objectively assessed biochemically by quantitating tamoxifen and AI drug and metabolite plasma concentrations as previously described.
Genotyping | Up to 18 months
  Germline deoxyribonucleic acid (DNA) will be genotyped by the University of Michigan Advanced Genomics Core using technology available at the time the analysis is performed

CONTACTS AND LOCATIONS:
Overall Officials: Norah L Henry, Principal Investigator — SWOG Cancer Research Network
Locations (490):
- United States (489):
  - Kingman Regional Medical Center, Kingman, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Marshall Cancer Center, Cameron Park, California
  - Mercy Cancer Center �� Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Epic Care-Dublin, Dublin, California
  - Kaiser Permanente Dublin, Dublin, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Saint John's Cancer Institute, Santa Monica, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Bayhealth Hospital Kent Campus, Dover, Delaware
  - Beebe South Coastal Health Campus, Frankford, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Bayhealth Hospital Sussex Campus, Milford, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Kaiser Permanente-Capitol Hill Medical Center, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Broward Health North, Deerfield Beach, Florida
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - The Watson Clinic, Lakeland, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - South Florida Baptist Hospital, Plant City, Florida
  - Tampa General Hospital, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northside Hospital - Duluth, Duluth, Georgia
  - Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Northside Hospital - Gwinnett, Lawrenceville, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Diagnostic Radiology Services LLC, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Straub Medical Center - Kahului Clinic, Kahului, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - The Queen's Medical Center - West Oahu, ‘Ewa Beach, Hawaii
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Advocate South Suburban Hospital, Hazel Crest, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Condell Memorial Hospital, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - West Suburban Medical Center, River Forest, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - HaysMed University of Kansas Health System, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Saint Joseph Mount Sterling, Mount Sterling, Kentucky
  - Louisiana State University Health Science Center, New Orleans, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Kaiser Permanente-Woodlawn Medical Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Kaiser Permanente-Gaithersburg Medical Center, Gaithersburg, Maryland
  - Kaiser Permanente - Kensington Medical Center, Kensington, Maryland
  - Kaiser Permanente - Largo Medical Center, Largo, Maryland
  - Kaiser Permanente Lutherville - Timonium Medical Center, Lutherville, Maryland
  - UM Saint Joseph Medical Center, Towson, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Lahey Medical Center-Peabody, Peabody, Massachusetts
  - Winchester Hospital, Winchester, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Academic Hematology Oncology Specialists, Grosse Pointe Woods, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Ascension Borgess Cancer Center, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Ascension Saint Mary's Hospital, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Ascension Saint Joseph Hospital, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - GenesisCare USA - Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pebble, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Las Vegas Urology - Pecos, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - GenesisCare USA - Las Vegas, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Las Vegas Prostate Cancer Center, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - GenesisCare USA - Vegas Tenaya, Las Vegas, Nevada
  - Las Vegas Urology - Cathedral Rock, Las Vegas, Nevada
  - Las Vegas Urology - Smoke Ranch, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - GenesisCare USA - Fort Apache, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - AtlantiCare Health Park-Cape May Court House, Cape May Court House, New Jersey
  - AtlantiCare Surgery Center, Egg Harbor, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Garnet Health Medical Center, Middletown, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Summa Health System - Akron Campus, Akron, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - Cleveland Clinic Mercy Hospital, Canton, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Summa Health Medina Medical Center, Medina, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Main Line Health Center-Collegeville, Collegeville, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Main Line Health Center-Exton, Exton, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Bryn Mawr Health Center, Newtown Square, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Phoenixville Hospital, Phoenixville, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - STCC at DHR Health Institute for Research and Development, Edinburg, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Kaiser Permanente-Burke Medical Center, Burke, Virginia
  - Centra Lynchburg Hematology-Oncology Clinic Inc, Lynchburg, Virginia
  - Kaiser Permanente Tysons Corner Medical Center, McLean, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Valley Medical Center, Renton, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Aurora Saint Luke's South Shore, Cudahy, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Marshfield Medical Center - Neillsville, Neillsville, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Ascension Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru

REFERENCES:
- [Derived] Henry NL, Unger JM, Vaidya R, Darke AK, Skaar TC, Fisch MJ, Hershman DL. Active symptom monitoring for premenopausal women with breast cancer initiating adjuvant endocrine therapy: Protocol for the SWOG S2010 randomized controlled efficacy trial. Contemp Clin Trials. 2024 Dec;147:107712. doi: 10.1016/j.cct.2024.107712. Epub 2024 Oct 10. PMID 39395534